CLINICAL TRIAL: NCT06828796
Title: Early Use of Tacrolimus in HLA-Mismatched Haploidentical Allogeneic Hematopoietic Transplantation With Post-Transplant Cyclophosphamide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1420
Record Dates: First submitted 2025-02-06; First posted 2025-02-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Disease and Disorders; Hematopoietic Cell Transplant
MeSH Terms: conditions — Hematologic Diseases; Disease | interventions — Tacrolimus; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tacrolimus + MMF + Post-Transplant Cyclophosphamide (Experimental): Cyclophosphamide 50mg/kg/d Days +3 and +4 after transplant Tacrolimus Day -1 to Day +90 or Day +180 after transplant MMF 15mg/kg PO TID Day 0 to Day +35
  Interventions: Drug: Tacrolimus; Drug: Cyclophosphamide; Drug: Mycofenolate mofetil

INTERVENTIONS:
Drug: Tacrolimus — Begins Day -1 and continues to Day +90 or Day +180 after transplant
Drug: Cyclophosphamide — Given Days +3 and +4 after transplant
Drug: Mycofenolate mofetil — Given Day 0 to Day +35 after transplant

SUMMARY:
To evalute the safety and efficacy in reducing Cytokine Release Syndrome after hematopoietic stem cell transplantation by introducing immunosuppression earlier in the transplant process

ELIGIBILITY:
Inclusion Criteria:

* Availability of a 5/10-8/10 mismatched (HLA-A, B, DR) haploidentical related donor with a negative HLA cross-match in the host vs. graft direction and willing to provide peripheral blood stem cells
* Karnofsky status >/= 70%
* Hematologic malignancy requiring allogeneic transplantation
* First allogeneic transplant only. Prior autologous transplant is allowed.

Exclusion Criteria:

* Poor cardiac function: LVEF <40%
* Poor pulmonary function: FEV1 and FVC <50% predicted
* Poor liver function: bilirubin >/= 3mg/dL (not due to hemolysis, Gilbert's or primary malignancy)
* Poor renal function: Creatinine >/= 2mg/dL or creatinine clearance (calculated or measured creatinine clearance is permitted) <40mL/min based on Traditional Cockcroft-Gault formula
* Women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* Patients who have any debilitating medical or psychiatric illness that would preclude their giving informed consent or their receiving optimal treatment and follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy in preventing CRS post transplant | 30 days
  Evaluate the incidence of CRS during the first 5 days following stem cell transplant by recording signs and symptoms based on CTCAE v5.0.

SECONDARY OUTCOMES:
Severity of CRS after stem cell transplant | 30 days
  Record incidence of CRS by grading signs and symptoms using the CTCAE v5.0, the day of onset of CRS, the duration of CRS, and admissions to the hospital for these events
Safety of administering early immunosuppression | 6 months
  Record incidence of acute graft-versus-host disease at 6 months by using the NIH Grading Consensus system
Safety of administering early immunosuppression | 1 year
  Record incidence of chronic graft-versus-host disease at 1 year by using the NIH Grading Consensus system

CONTACTS AND LOCATIONS:
Overall Officials: Melhem Solh, MD, Principal Investigator — The Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the trial will be shared on clinicaltrials.gov
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] Solh MM, Dickhaus E, Solomon SR, Morris LE, Zhang X, Holland HK, Bashey A. Fevers post infusion of T-cell replete hla mismatched haploidentical hematopoietic stem cells with post-transplant cyclophosphamide: risk factors and impact on transplant outcomes. Bone Marrow Transplant. 2019 Nov;54(11):1756-1763. doi: 10.1038/s41409-019-0522-4. Epub 2019 Apr 5. PMID 30953027
- [Result] Tang J, Jensen RR, Bryan B, Hoda D, Hunter BD. Reduced Cytokine Release Syndrome and Improved Outcomes with Earlier Immunosuppressive Therapy in Haploidentical Stem Cell Transplantation. Transplant Cell Ther. 2024 Apr;30(4):438.e1-438.e11. doi: 10.1016/j.jtct.2024.01.076. Epub 2024 Jan 26. PMID 38281591
- [Result] Abboud R, Wan F, Mariotti J, Arango M, Castagna L, Romee R, Hamadani M, Chhabra S. Cytokine release syndrome after haploidentical hematopoietic cell transplantation: an international multicenter analysis. Bone Marrow Transplant. 2021 Nov;56(11):2763-2770. doi: 10.1038/s41409-021-01403-w. Epub 2021 Jul 14. PMID 34262142
- [Result] Abboud R, Keller J, Slade M, DiPersio JF, Westervelt P, Rettig MP, Meier S, Fehniger TA, Abboud CN, Uy GL, Vij R, Trinkaus KM, Schroeder MA, Romee R. Severe Cytokine-Release Syndrome after T Cell-Replete Peripheral Blood Haploidentical Donor Transplantation Is Associated with Poor Survival and Anti-IL-6 Therapy Is Safe and Well Tolerated. Biol Blood Marrow Transplant. 2016 Oct;22(10):1851-1860. doi: 10.1016/j.bbmt.2016.06.010. Epub 2016 Jun 16. PMID 27318038
- [Result] Ruggeri A, Labopin M, Battipaglia G, Chiusolo P, Tischer J, Diez-Martin JL, Bruno B, Castagna L, Moiseev IS, Vitek A, Rovira M, Ciceri F, Bacigalupo A, Nagler A, Mohty M. Timing of Post-Transplantation Cyclophosphamide Administration in Haploidentical Transplantation: A Comparative Study on Behalf of the Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2020 Oct;26(10):1915-1922. doi: 10.1016/j.bbmt.2020.06.026. Epub 2020 Jul 6. PMID 32645444
- [Result] Chiusolo P, Bug G, Olivieri A, Brune M, Mordini N, Alessandrino PE, Dominietto A, Raiola AM, Di Grazia C, Gualandi F, Van Lint MT, Ferrara F, Finizio O, Angelucci E, Bacigalupo A. A Modified Post-Transplant Cyclophosphamide Regimen, for Unmanipulated Haploidentical Marrow Transplantation, in Acute Myeloid Leukemia: A Multicenter Study. Biol Blood Marrow Transplant. 2018 Jun;24(6):1243-1249. doi: 10.1016/j.bbmt.2018.01.031. Epub 2018 Feb 5. PMID 29421292
- [Result] Bashey A, Zhang X, Sizemore CA, Manion K, Brown S, Holland HK, Morris LE, Solomon SR. T-cell-replete HLA-haploidentical hematopoietic transplantation for hematologic malignancies using post-transplantation cyclophosphamide results in outcomes equivalent to those of contemporaneous HLA-matched related and unrelated donor transplantation. J Clin Oncol. 2013 Apr 1;31(10):1310-6. doi: 10.1200/JCO.2012.44.3523. Epub 2013 Feb 19. PMID 23423745
- [Result] Mayumi H, Umesue M, Nomoto K. Cyclophosphamide-induced immunological tolerance: an overview. Immunobiology. 1996 Jul;195(2):129-39. doi: 10.1016/S0171-2985(96)80033-7. PMID 8877390
- [Result] Jones RJ, Barber JP, Vala MS, Collector MI, Kaufmann SH, Ludeman SM, Colvin OM, Hilton J. Assessment of aldehyde dehydrogenase in viable cells. Blood. 1995 May 15;85(10):2742-6. PMID 7742535
- [Result] Fuchs EJ. Haploidentical transplantation for hematologic malignancies: where do we stand? Hematology Am Soc Hematol Educ Program. 2012;2012:230-6. doi: 10.1182/asheducation-2012.1.230. PMID 23233586